CLINICAL TRIAL: NCT01630655
Title: An Open Label, Randomised, 2-period, 2-treatment, 2-sequence, Cross-over, Single-dose Bioequivalence Study of Felodipine Extended-Release Tablets USP 10 mg (Test, Torrent Pharmaceuticals Ltd., India) Versus Felodipine Extended-Release Tablets USP 10 mg (Reference, Mylan Pharmaceuticals Inc., USA) in Healthy Human Volunteers Under Fasting Condition
Brief Title: Bioequivalence Study of Torrent Pharmaceuticals Ltd's Felodipine Extended-Release Tablets Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 426-09
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Torrent's Felodipine Extended-Release Tablets

SUMMARY:
Objective:

Primary objective of the present study was to compare the single dose bioavailability of Torrent's Felodipine Extended-Release Tablets USP 10 mg and Innovator's (Mylan Pharmaceuticals Inc., USA) Felodipine Extended-Release Tablets USP 10 mg. Dosing periods were separated by a washout period of 17 days during fasting study.

Study Design:

Open-Label, Randomised, two Period, two treatment, Crossover, Single-Dose Bioequivalence Study

ELIGIBILITY:
Inclusion Criteria:

* Healthy males within the age range of 18 to 50 years.
* A body mass index within 18-25 Kg/m2.
* Given written informed consent to participate in the study.
* Absence of diseases markers of HIV 1 & 2, Hepatitis B & C virus and RPR.
* Absence of significant disease or clinically significant abnormal laboratory
* values on laboratory evaluation, medical history and physical examination during the screening.
* A normal 12-lead ECG.
* A normal chest X-Ray.
* Comprehension of the nature and purpose of the study and compliance with the requirements of the entire protocol.
* No history or no evidence of hypersensitivity or idiosyncratic reactions to other nitrates or nitrites.
* No history of allergic rash.
* No history of significant systemic diseases.
* No history of psychiatric disorders or addiction to any recreational drug or drug dependence.
* No donation of blood within 56 days prior to study check-in.
* No participation in any clinical study within the past 56 days.
* No receipt of any prescription drugs or OTC products, with in two weeks prior to study check-in.
* No history of dehydration from diarrhea, vomiting or any other reason within a period of 24 hours prior to study check-in.
* No family history of neurological disorders.
* Not consumed alcohol and xanthine containing food and beverages, cigarettes and tobacco products, for at-list 48 hours, prior to study check-in.
* Negative results for drugs of abuse in urine and alcohol breath analysis during check-in of each period.
* Not consumed grape fruit juice within the 48 hours prior to study check-in.

Exclusion Criteria:

* Blood pressure Systolic> 140 mm Hg and < 110 mm Hg Diastolic< 70 mm Hg > 90 mm Hg
* History of seizures
* History of alcohol consumption for more than 2 units/day.
* High caffeine or tobacco consumption
* History of difficulty with donating blood or difficulty in accessibility of veins.
* Any unusual or abnormal diet, for whatever reason e.g. fasting due to religious reasons.
* Used any pharmacological agents known to significantly induce or inhibit drug metabolizing enzymes within 14 days of the start of the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult

PRIMARY OUTCOMES:
bioequivalence based on Composite of Pharmacokinetics
  bioequivalence; 90% geometric confidence interval of the ratio of least-squares means of the test to reference product should be within 80.00% - 125.00% for AUC-unf, AUCo-t and Cmax.

CONTACTS AND LOCATIONS:
Locations (1):
- AXIS Clinicals Limited(formerly Trident Life Sciences Ltd.), Miyāpur, Hyderabad, India